CLINICAL TRIAL: NCT02837393
Title: Understanding the Urine Electrolyte Profile of the Individual Renal Unit
Status: Terminated | Type: Observational
Why Stopped: Low Recruitment and Enrollment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00099408
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Kidney Calculi; Nephrolithiasis; Urolithiasis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urolithiasis | interventions — Urinary Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- History of Kidney Stones: Participants with a history of kidney stones who will be undergoing kidney surgery.
  Interventions: Procedure: Ureteral catheterization
- No History of Kidney Stones: Participants without a history of kidney stones who will be undergoing kidney surgery.
  Interventions: Procedure: Ureteral catheterization

INTERVENTIONS:
Procedure: Ureteral catheterization — During ureteral catheterization, urine samples will be obtain from each kidney

SUMMARY:
The investigators objective is to determine if urinary electrolyte abnormalities exist in only one or both kidneys in participants with and without a history of kidney stones. To meet this objective, the investigators are going to take urine samples from each kidney at the time of kidney stone surgery. The samples will then be analyzed for absolute and relative differences in the concentrations of urine electrolytes, such as calcium.

DETAILED DESCRIPTION:
Nephrolithiasis is common within the general population. Although the majority of patients with a symptomatic stone event will not require surgical intervention, the rate of recurrence is high. Therefore, reducing this rate of recurrence is important.

Traditionally, this has been achieved with a combination of serum and urine metabolic evaluation followed by targeted medication and dietary interventions. Specifically, it is recommended that a single 24-hour urine collection for analysis of urine electrolytes be performed. A 24-hour urine collection is bladder urine, which is pooled urine from both kidneys. The urine is then analyzed for the relative and absolute concentrations of electrolytes and small molecules known to be associated with stone formation. These include creatinine, calcium, citrate, oxalate, potassium, magnesium, phosphate, uric acid, and urate.

When an abnormality is detected on a 24-hour urine collection the assumption is that this is due to a global metabolic defect present in both kidneys. However, this may not be the case. It is possible there could be a relative imbalance with both kidneys having a defect, but to different degrees (or different defects in one or multiple electrolytes). It is also possible that one kidney has a dominant defect, but the contralateral kidney is normal, and therefore the 24-hour urine collection would only represent the dominant kidney with the defect. Finally, it is possible that the converse is true. One kidney has no defect, but the contralateral kidney has a minor defect. In this example, the 24-hour urine collection would appear normal as the dominant normal kidney masks the minor defect. This concept of differential kidney electrolyte handling was previously described in children. Therefore, understanding individual kidney metabolic profiles is important.

The purpose of the investigators' study will be to (1) characterize the urine electrolyte profile of each individual renal unit; (2) identify participants who have differences between their renal unit urine electrolyte profiles, and their renal units and bladder urine electrolyte profiles; and (3) correlate differences in renal unit urine electrolyte profiles with clinical manifestations of kidney stones, such as stone formation or growth. By characterizing individual renal unit urine electrolyte profiles, the investigators' may be able to isolate a phenotype of stone formers who would not otherwise be identified with traditional 24-hour urine collection. The investigators' can then target this phenotype in future investigations with dietary and medication interventions to hopefully prevent future stone events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Planed upper urinary tract surgery for a diagnosis of nephrolithiasis, hematuria, ureteral stricture, ureteropelvic junction obstruction, hydronephrosis, or intra-operative identification of the ureters.

Exclusion Criteria:

1. History of an anatomic abnormality of the urinary tract.
2. History of a solitary kidney.
3. Untreated or a history of lower or upper urinary tract urothelial malignancy.
4. Active urinary tract infection.
5. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be a prospective cohort study conducted within the Department of Urology at Johns Hopkins Hospital and Bayview Medical Center. The study population will be comprised of a convenience sample of participants 18 years of age or older who will be undergoing upper urinary tract surgery as part of routine clinical care for a diagnosis of nephrolithiasis, hematuria, ureteral stricture, ureteropelvic junction obstruction, hydronephrosis, or intra-operative identification of the ureters.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Concentrations of urine electrolytes | 1 year
  The investigators' will determine if there is a difference in urine electrolyte concentrations within individuals between the two kidneys, and across individuals in those with and without a history of kidney stones.

CONTACTS AND LOCATIONS:
Overall Officials: Justin B Ziemba, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No